CLINICAL TRIAL: NCT06884800
Title: Laparoscopic Toupet's Fundoplication: Is it Proper Solution of Radiological Negative, Endoscopically Positive Hiatal Hernia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Salah, Lecturer of General Surgery, Faculty of Medicine, Minia University, Minia, Egypt., Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1241/08/2024
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Laparoscopic Toupet Fundoplication; Radiological Negative; Endoscope; Hiatal Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic toupet fundoplication group (Experimental): Patients will undergo laparoscopic toupet fundoplication.
  Interventions: Procedure: Laparoscopic toupet fundoplication

INTERVENTIONS:
Procedure: Laparoscopic toupet fundoplication — Patients will undergo laparoscopic toupet fundoplication.

SUMMARY:
This study aims to assess the feasibility and effectiveness of laparoscopic toupet fundoplication (LTF) for treating gastroesophageal reflux disease (GERD) symptoms and disease-specific Quality of Life (QoL).

DETAILED DESCRIPTION:
Heartburn, regurgitation, dysphagia, and chest pain are regarded as common esophageal symptoms of gastroesophageal reflux disease (GERD). On the other hand, there are very few reports of laryngopharyngeal reflux (LPR), which is associated with persistent upper airway contact, acidic and non-acidic reflux, and aerosol that results in posterior laryngitis, edema, and glottis erythema.

Proton-pump inhibitor (PPI) therapy, Laparoscopic Nissen Fundoplication (LNF), and Laparoscopic Toupet Fundoplication (LTF) have been proven to be effective for the treatment of GERD. However, the therapeutic management of patients with hiatal hernia is debated and treatment remains empirical. Previous studies on PPI therapy and LNF had been published with promising but controversial results. Therefore, the role of LTF is even less explored and evidence is scarce

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old.
* Both sexes.
* Hiatal hernia patients (Hill's grade III & IV) by endoscopy and negative by radiology indicated for Toupet fundoplication.

Exclusion Criteria:

* Recurrent patients.
* Age above 70 years old
* Unfit for surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of recurrence | 1 year postoperatively
  Incidence of recurrence will be recorded

SECONDARY OUTCOMES:
Incidence of anatomical failure | 1 year postoperatively
  Incidence of anatomical failure will be recorded
Incidence of complications | 1 year postoperatively
  Incidence of complications such as dysphagia, chest pain on eating, gas-bloat, postprandial fullness, restriction in belching, and increased flatus will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author